CLINICAL TRIAL: NCT01025037
Title: A Prospective, Multi-Center, Single-Arm Study to Assess Clinical Outcomes In Primary Open or Mini-Open Rotator Cuff Repair Using Conexa Graft Reinforcement
Brief Title: Outcomes in Rotator Cuff Repair Using Graft Reinforcement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Trauma and Extremities (Industry)
Collaborators: LifeCell (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tornier-LIFC LFC2008.03.02
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator Cuff Tear, Large, Massive, Rotator, Cuff. Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Conexa Reconstructive Tissue Matrix (Other): Conexa will be placed as a soft tissue reinforcement at the rotator cuff repair site
  Interventions: Device: Conexa Reconstructive Tissue Matrix

INTERVENTIONS:
Device: Conexa Reconstructive Tissue Matrix — Conexa will be placed as a soft tissue reinforcement in primary open or mini-open rotator cuff repair procedures
  Other Names: Conexa, Conexa TM

SUMMARY:
The purpose of this study is to evaluate patient shoulder functional outcomes following rotator cuff repairs reinforced with a surgical mesh.

DETAILED DESCRIPTION:
Conexa is a surgical mesh derived from porcine dermis and processed to produce an acellular dermal matrix. It is designed to perform as a surgical mesh for use as a soft tissue patch to reinforce soft tissue where weaknesses exist and for the surgical repair of damaged or ruptured soft tissue membranes. The purpose of this post-market clinical study is to collect safety and efficacy data when Conexa is used to repair torn tendons of the rotator cuff. Conexa will be used in accordance with its labeling for this clinical study.

ELIGIBILITY:
Inclusion Criteria:

The patient:

1. is an adult male or female between the ages of 40-70 years old;
2. has repairable primary large retracted two-tendon rotator cuff tears measuring from 3 cm to 5 cm;
3. requires surgical repair of single rotator cuff (i.e. one limb);
4. has movement of the non-operative arm defined as shoulder elevation of equal to or greater than 90 degrees and is able to perform postoperative exercises;
5. is able to return for all scheduled and required study visits;
6. is able to provide written informed consent for study participation.

Exclusion Criteria:

The patient:

1. has irreparable large rotator cuff tears that are found intra-operatively. Note: irreparable is defined by the inability to approximate the tendon to the tuberosity without tension;
2. has a rotator cuff tear < 3cm (measured intra-operatively);
3. has a rotator cuff tear > 5cm (measured intra-operatively);
4. has a rotator cuff tear where the subscapularis tendon is disrupted/requires repair;
5. has grade 3 or 4 fatty infiltration of the rotator cuff;
6. has had prior surgical repair to the affected shoulder;
7. is American Society of Anesthesiologists (ASA) Class 4 or 5 (See Appendix I);
8. is a tobacco user; unless tobacco free 6 months prior to surgery and willing to remain tobacco free for the duration of the study.
9. has lower limb injuries requiring walking assist devices such as crutches and walkers;
10. has a known collagen disorder, including systemic lupus erythematous (SLE), rheumatoid arthritis (RA), polymyositis, scleroderma, ankylosing spondylitis, dermatomyositis, osteogenesis imperfecta or the inherited disorders of Sjogren, Larsen, Raynaud, Ehlers-Danlos or Marfan syndrome.
11. has obstacles that pose an inordinately high surgical risk, in the judgment of the certified surgeon;
12. has co-morbid factors which predispose to postoperative infection, such as insulin dependent diabetes, chronic steroid use, malnourishment, cancer, or co-existent infection;
13. has a history of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or drug abuse or addiction;
14. is enrolled or plans to enroll in another clinical trial during this study that would affect the patient's safety or results of this trial;
15. has any of the conditions identified within the labeled contraindications, i.e. sensitivity to porcine derived products or polysorbate.
16. has an inability to have a closed MRI conducted.
17. needs a re-operation for a re-tear of the rotator cuff.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-10; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Iannotti, MD, Study Director — Cleveland, OH; John Sperling, MD, Study Director — Rochester, MN
Locations (6):
- United States (6):
  - Orthopaedic Clinical Association, Phoenix, Arizona
  - Rush University Medical Center, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - OrthoNeuro, New Albany, Ohio
  - Rotheman Institute, Philadelphia, Pennsylvania
  - West Virginia University, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Conexa: Rotator cuff repair using Conexa
Period: Overall Study
Arm/Group | Conexa
Started | 61
Completed | 50
Not Completed | 11
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Conexa
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 38
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 5
  White | 56
Region of Enrollment [Number; unit: participants]
  United States | 61
Height [Mean (Standard Deviation); unit: cm] | 171.5 (11.3)
Weight [Mean (Standard Deviation); unit: kg] | 94.9 (24.9)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: American Shoulder and Elbow Score (ASES)
Description: The ASES evaluation generally has a patient self-evaluation section and a physician assessment section. The patient self-evaluation section of the form contains visual analog scales for pain, instability, an activities of daily living (ADL) questionnaire. The physician assessment section includes an area to collect demographic information and assesses range of motion, specific physical signs, strength, and stability. A shoulder score can be derived from the visual analogue scale score for pain (50%) and the cumulative activities of daily living score (50%) (Richards, Bigliani, Gartsman, Iannotti, & Zuckerman, 1994). The ASES evaluation has a total of 100 points possible; with 100 being the best possible outcome, and 0 being the worst.
Time Frame: baseline, post-op months 3, 6, 12, and 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conexa
Number analyzed (Participants) | 61
units on a scale
  Baseline Measurement | 48.7 (20.2)
  3 Month Measurement | 69.4 (16.2)
  6 Month Measurement | 79.9 (17.7)
  12 Month Measurement | 85.4 (18.4)
  24 Month Measurement | 90.4 (15.3)

2. Secondary Outcome: Rotator Cuff Re-tear Evaluation
Description: Subjects will have MRI to assess healing of the repaired tendon at 6 and 12 months post-op. The rate of re-tear will be reported.
  Two different definitions of a re-tear were used for the analysis.
  1. Primary definition (used for analysis of the secondary objective): Full thickness tear that is 80% or greater in length of the original tear size.
  2. Sub-analysis: Full thickness tear one centimeter or greater in length.
Time Frame: Post-op months 6 and 12
Population: Participants were analyzed at 6 and 12 months post-op. 2 participants not analyzed due to exclusion prior to 6 month post op visit.
Measure: Number; unit: percentage of participants
Arm/Group | Conexa
Number analyzed (Participants) | 59
percentage of participants
  80% re-tear Definition, 6 months | 18.5
  80% re-tear definition, 12 months | 16.9
  1 cm re-tear definition, 6 months | 32.2
  1 cm re-tear definition, 12 months | 33.9

3. Other Pre Specified Outcome: Incidence of Complications, Including Infection
Description: Complications were summarized by reporting adverse events of special interest. AEs of special interest were defined as any reported infection (incision, wound, surgical site), seroma, hematoma, inflammation (surgical site, wound), and re-tear. The re-tear rate reported in this section is the number reported via AE or surgical intervention (not the MRI results). The AEs of special interest were chosen because they are in alignment with the potential complications listed on the product insert.
Time Frame: All time points
Measure: Number; unit: percentage of participants
Arm/Group | Conexa
Number analyzed (Participants) | 61
percentage of participants
  Inflammation (surgical site, wound);Severity: Mild | 9.8
  Re-tear;Severity: Mild | 9.8

4. Primary Outcome: Adjusted Constant-Murley Score
Description: The Constant-Murley Shoulder Score is a 100-point functional shoulder assessment tool in which higher scores reflect increased function. The subjective variables are pain (15 points) and function (Activities of Daily Living - sleep, work, recreation/sport) (20 points), for a total of 35 points. The objective variables are active range of motion (clinician assessment) (40 points) and strength (25 points), for a total of 65 points (Stiller & Uhl, 2005).
Time Frame: baseline, post-op months 6, 12, and 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conexa
Number analyzed (Participants) | 61
units on a scale
  Baseline Measurement | 45.4 (15.2)
  6 Month Measurement | 62.9 (11.6)
  12 Month Measurement | 68.7 (11.3)
  24 Month Measurement | 71.7 (9.6)

5. Primary Outcome: Simple Shoulder Test (SST)
Description: The Simple Shoulder Test (SST): a series of 12 "yes" or "no" questions the patient answers about the function of the involved shoulder; 2 questions relate to pain, 7 questions relate to function and 3 questions relate to range of motion. The answers to these questions (yes = 1, no = 0) provides a standardized way of recording the function of a shoulder before and after treatment (McClure & Michener, 2003). A score of 12 on the Simple Shoulder test represents the best possible outcome, while a score of 0 represents the worst possible outcome.
Time Frame: baseline, post-op months 3, 6, 12, and 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conexa
Number analyzed (Participants) | 61
units on a scale
  Baseline Measurement | 5.0 (2.6)
  3 Month Measurement | 6.4 (3.0)
  6 Month Measurement | 8.7 (2.7)
  12 Month Measurement | 9.9 (2.5)
  24 Month Measurement | 10.6 (2.2)

6. Secondary Outcome: Isometric Strength
Time Frame: baseline, post-op months 6, 12, and 24
Measure: Mean (Standard Deviation); unit: newtons (N)
Arm/Group | Conexa
Number analyzed (Participants) | 61
newtons (N)
  Baseline Measurement | 34.4 (26.8)
  6 Month Measurement | 61.9 (52.8)
  12 Month Measurement | 83.0 (71.7)
  24 Month Measurement | 78.6 (63.2)

ADVERSE EVENTS:
Arm/Group | Conexa
Serious Adverse Events (participants affected / at risk) | 1/61
Other Adverse Events (participants affected / at risk) | 35/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conexa (N=61)
Wound Infection (Infections and infestations) | 1 — Subject underwent irrigation and debridement of the shoulder, was given antibiotics, and the SAE was resolved without sequelae.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conexa (N=61)
Mild Rotator Cuff Syndrome (Injury, poisoning and procedural complications) | 8
Moderate Rotator Cuff Syndrome (Injury, poisoning and procedural complications) | 5
Mild Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 10
Mild Inflammation (surgical site, wound) (Musculoskeletal and connective tissue disorders) | 6
Re-Tear (Musculoskeletal and connective tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less